CLINICAL TRIAL: NCT07180108
Title: PRoMiSS: Psilocybin and the Role of Music in Set and Setting
Acronym: PRoMiSS
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00372917
Record Dates: First submitted 2025-09-02; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Psilocybin; Music Intervention
Keywords: Psilocybin; Set and Setting; Music Cognition; Music-evoked autobiographical memory; Emotion; Altered State of Consciousness; Psychedelics; Memory
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: open-label psilocybin (25mg) but music condition is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 6 hour playlist of music (Experimental): A 6 hour playlist of music.
  Interventions: Drug: Psilocybin (high dose); Behavioral: Playlist 1; Behavioral: Playlist 2; Behavioral: Playlist 3; Behavioral: Playlist 4; Behavioral: Playlist 5

INTERVENTIONS:
Drug: Psilocybin (high dose) — 25 mg pill
  Other Names: DMF#037635 (Type II); Purisys LLC; Psilocybin Drug Substance
Behavioral: Playlist 1 — Six hour playlist
Behavioral: Playlist 2 — A six hour playlist
Behavioral: Playlist 3 — A six hour playlist
Behavioral: Playlist 4 — A six hour playlist
Behavioral: Playlist 5 — A six hour playlist

SUMMARY:
The goal of this clinical trial is to understand how personally meaningful, autobiographically salient music compares to standardized playlists when combined with psilocybin in healthy adults ages 21 to 75. The main questions it aims to answer are:

Does autobiographically salient music lead to stronger emotional responses to music, greater acute subjective effects, and more lasting improvements in mood, affect, and well-being compared to standardized or ambient playlists?

How are brain and body responses - including EEG activity, respiration, heart rate, and skin conductance - influenced by autobiographically salient music under psilocybin?

Do brain and body responses to specific music features differ when the music is autobiographically salient compared to non-salient playlists?

Researchers will compare five music conditions: three conditions where an 80-minute block of autobiographically salient music is placed at different points in the 6-hour psilocybin session (0-80 minutes, 80-160 minutes, or 240-320 minutes), a standardized Johns Hopkins psilocybin playlist, and an ambient playlist with no autobiographical content.

Participants will:

* Take a single oral dose of psilocybin (25 mg) during one study session
* Listen to one of the five music conditions while reclining in a comfortable setting
* Complete questionnaires about emotions, acute, subjective effects, insight, etc.
* Undergo EEG and physiological monitoring (respiration, heart rate, skin conductance) during the session
* Complete MRI brain scans before the session and 1 week after psilocybin
* Return for follow-ups at 1 day, 1 week, and 1 month after psilocybin
* At 1 month, complete a qualitative interview and a nondrug EEG music listening session, where the participant's hear either music from the participant's own psilocybin session or music from another participant's session

DETAILED DESCRIPTION:
Classic psychedelics such as psilocybin reliably alter consciousness, producing changes in perception, emotion, and meaning-making. Music has long been recognized as an important component of psychedelic therapy, serving to guide the experience and shape its trajectory. However, little is known about how different types of music influence outcomes, particularly music that is personally meaningful to participants.

This study will investigate the effects of autobiographically salient (AS) music compared to standardized playlists during high-dose psilocybin sessions. The goal is to understand how personally relevant music modulates acute subjective experiences, emotional responses, and longer-term psychological outcomes. In addition, the study will examine brain and body responses to music under psilocybin, including how these responses differ when music is autobiographically salient.

The central questions are whether AS music enhances emotional depth, psychological insight, and well-being more than non-autobiographical playlists, and whether the timing of AS music during the session influences these effects. Participants will be followed up after the psilocybin session to assess both short-term and longer-term outcomes, including well-being, mood, and meaning-making.

This trial represents one of the first controlled investigations into how personalized music contributes to the therapeutic potential of psychedelics. Findings may help optimize music-based interventions in psychedelic therapy and improve understanding of the role of music in shaping altered states of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* • Fluent in English

  * No hearing impairment
  * Right-handed
  * Have a screening weight ≥ 40 kg (88.18 lbs) with BMI ≥16.
  * Be medically stable as determined by screening for medical problems via a personal interview, a medical history, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
  * Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
  * Agree to refrain from using any psychoactive drugs within 24 hours of each drug administration. The exceptions are caffeine and nicotine, which can be consumed before arriving for drug administration sessions.
  * Agree not to take any as needed (PRN) medications on the mornings of drug sessions
  * Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
  * Agree not to use any hair conditioner 24-hours before EEG sessions (Visits 3, 4, and 7)
  * Females of child-bearing potential must agree to use highly effective methods of contraception (defined as use of an intrauterine device, vaginal ring, or implanted or oral hormonal contraceptives) during the study
  * Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti- inflammatory drugs, and common doses of vitamins and minerals.
  * Have limited lifetime use of hallucinogens, if any (the following criteria are preferred: no use in the past 5 years; total hallucinogen use less than 10 times)
  * Proof of COVID-19 vaccination.

Exclusion Criteria:

* • Unusually low reward response to music (defined as a majority of responses of "1" on the BMRQ)

  * Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing highly effective means of contraception
  * Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged corrected QT interval (QTc) interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack (TIA) in the past year
  * Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
  * Currently taking psychoactive prescription medication on a regular (e.g., daily) basis - exceptions may be made at the discretion of the study team physician for participants taking medications with short half-life if participants are able to abstain from taking the medication during session days (e.g. methylphenidate taken for attention or hyperactivity)
  * Currently taking on a regular (e.g., daily) basis any medications that have a primary centrally-acting serotonergic effect, including Monoamine Oxidase Inhibitors (MAOIs). For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
  * Current or past history of meeting Diagnostic and Statistical Manual (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I Disorder
  * Current or history within one year of meeting DSM-5 criteria for a moderate or severe substance use disorder. If a nicotine user, consuming the equivalent of more than 10 cigarettes per day.
  * Have a first-degree relative with schizophrenia spectrum or other psychotic disorders, or bipolar disorder with mania (except substance/medication-induced or due to another medical condition)
  * Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
  * History of a medically significant suicide attempt as assessed by a study team clinician
  * Standard MRI contraindications: head trauma, claustrophobia incompatible with scanning, contraindicated medical devices, prior history as a metal worker and/or certain metallic objects in the body -- must complete MRI screening form and be approved by MRI technologist before each scan
  * History of migraine.
  * History of angiotensin-converting enzyme inhibitor (ACEi) angioedema

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Challenging Experiences Questionnaire | Immediately at the end of their experimental session
  The Challenging Experience Questionnaire (CEQ) is a self-report measure designed to assess the intensity and quality of difficult or distressing experiences during psychedelic states.
  Zero is equivalent to no challenging experiences and 5 is an extreme (more than ever before in my life). Higher CEQ = "more difficult." That's generally worse for safety and usually not what predicts the best clinical gains.
Psychological Insight Questionnaire (PIQ) | Immediately at end of experimental session
  The Psychological Insight Questionnaire (PIQ) is a validated self-report measure developed to assess psychological insight experiences following a psychedelic session. It was designed to capture the extent to which individuals gain meaningful self-related or therapeutic insights during and after acute psychedelic states.
  The PIQ is scored 0 (not at all) to 6 Extremely (more than ever before in my life). A higher score is associated with better outcomes.
Core Flow State Scale (C-FSS) | Immediately at end of experimental session
  The Core Flow State Scale (CFSS) is a validated self-report measure designed to assess the subjective experience of flow, the psychological state of deep absorption, enjoyment, and optimal engagement in an activity.
  The CFSS is scored from 1 (Strongly Disagree) to 5 (Strongly Agree). A higher score is better.
Mystical Experiences Questionnaire (MEQ-30) | Immediately at end of experimental session
  The Mystical Experience Questionnaire (MEQ) is the most widely used measure for assessing the phenomenological features of mystical-type experiences occasioned by psychedelics.
  The MEQ is measured from 0 (not at all) to 5 extreme (ore than ever before in my life and stronger than 4). A higher MEQ score is associated with better outcomes.
Experience of Unity (11D-ASC) | Immediately after experimental session
  A sense of oneness with the environment or the universe, dissolving boundaries between self and world.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Experience of Unity scores are generally better
Change in EEG oscillatory power across canonical frequency bands (µV²/Hz) | During experimental session up to 10 hours
  EEG - spectral analysis - Electroencephalography (EEG) is a non-invasive neuroimaging method that measures the brain's electrical activity via electrodes placed on the scalp.
  Change in EEG oscillatory power across canonical frequency bands (delta, theta, alpha, beta, gamma) during music listening under psilocybin. Analyses will be conducted at the scalp sensor level using Statistical Parametric Mapping, version 12 (SPM12).
  Group-level contrasts of oscillatory power changes (µV²/Hz) across music conditions
Music Ratings: Autobiographical Salience | 1-day following experimental session and immediately post 1-month EEG music listening session
  Ratings of autobiographical salience for each song. Autobiographical salience is scored from 0 (none) to 4 (extremely autobiographically salient). More autobiographically salient music is thought to be better.
Spiritual Experience - Altered States of Consciousness (ASC-11D) | Immediately after experimental session
  Feelings of sacredness, transcendence, or contact with a higher reality.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Spiritual Experience scores are generally better.
Blissful State (11D-ASC) | Immediately after experimental session
  Intense feelings of happiness, peace, and contentment.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Blissful State scores are generally better.
Insightfulness (11D-ASC) | Immediately after experimental session
  Deep personal or existential insights, perceived understanding of self or reality.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Insightfulness scores are generally better.
Disembodiment (11D-ASC) | Immediately after experimental session
  Altered sense of the body, including floating, detachment, or out-of-body experiences.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Disembodiment scores are generally neutral or ambivalent. Mild forms may support ego dissolution and positive outcomes, but extreme disembodiment sometimes predicts challenging experiences.
Impaired Cognition & Control (11D ASC) | Immediately after experimental session
  Difficulty thinking clearly, controlling thoughts, or performing tasks.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Impaired Cognition and Control are generally linked with confusion and less therapeutic benefit.
Anxiety (11D-ASC) | Immediately after experimental session
  Fear, unease, or paranoid thoughts during the experience.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Higher Anxiety is generally linked with lower acute well-being, though may sometimes precede later benefit if well-supported.
Complex Imagery (11D-ASC) | Immediately after experimental session
  Vivid, detailed visual imagery of objects, scenes, or entities.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Complex Imagery is generally neutral. Vivid imagery contributes to meaningfulness but is not a consistent predictor of therapeutic change.
Elementary Imagery (11D-ASC) | Immediately after experimental session
  Simple visual patterns such as colors, shapes, or geometric forms.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Elementary Imagery is generally neutral. It is a common perceptual effect of psilocybin but is not strongly tied to long-term outcomes.
Audio-Visual Synesthesia (11D-ASC) | Immediately after experimental session
  Cross-modal experiences, such as hearing colors or seeing sounds.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Audio-Visual Synesthesia is generally neutral. It is an interesting phenomenology, but has weak association with outcomes.
Changed Meaning of Percepts (11D-ASC) | Immediately after experimental session
  Altered interpretation of ordinary sensory stimuli, often with symbolic or novel significance.
  The 11D-ASC is a self-report questionnaire designed to assess the phenomenology of altered states of consciousness induced by psychedelics and other methods (e.g., meditation, sensory deprivation). There are 11 dimensions.
  Questions are scored from 0 (No, not more than usual) to 100 (Yes, much more than usual). Changed Meaning of Percepts can be positive or negative. It can enhance therapeutic meaning and insight (positive), but in some cases may drive paranoia or misinterpretation (negative).

SECONDARY OUTCOMES:
Brain Activity measured by Blood Oxygenation Level Dependent signal | At Preparation Session 2 (before experimental session) and 1-week post experimental session
  Functional Magnetic Resonance Imaging (fMRI) is a non-invasive neuroimaging technique that measures brain activity by detecting changes in blood oxygenation (BOLD signal), which reflects local neural activity.
  We will be measuring a change in BOLD signal between the pre-experiment (preparation 2) and 1-week post-experiment. The main contrasts will include:
  * Pre vs Post (all music)
  * Pre vs Post (Autobiographically Salient music)
  * Pre vs. Post (JHC playlist music)
  * Pre vs Post (AMB playlist music)
Joyful Activation (GEMS-Joy) | 1-day after experimental session
  Cheerfulness, enthusiasm, vitality, dancing or movement impulses
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  A higher Joyful Activation score is generally positive and liked to pleasurable absorption and well-being.
Trait Impulsivity Questionnaire (BIS-11) | Preparation (pre experiment), 1-week post experimental session, and 1-month post experimental session
  The Barratt Impulsiveness Scale (BIS-11) is one of the most widely used self-report instruments for assessing trait impulsivity.
  The BIS-11 is scored from 0 (Rarely/Never) to 3 (Almost Always/Always). Generally lower impulsivity is better.
Core Dispositional Flow Scale (C DFS) | Preparation (pre experiment), 1-week post experimental session, and 1-month post post experimental session
  The Core Dispositional Flow Scale (CDFS) is a brief, validated self-report instrument designed to measure an individual's general tendency to experience flow across activities and contexts.
  The CDFS is measured from 1 (never) to 5 (always). A higher score is generally better.
Satisfaction With Life Scale (SWLS) | Preparation (baseline), 1-week post experimental session , and 1-month post experimental session
  The Satisfaction With Life Scale (SWLS) is a brief self-report instrument designed to measure global cognitive judgments of one's overall life satisfaction.
  The SWLS is measured from 1 (strongly disagree) to 7 (strongly agree). A higher score is better.
Big Five Inventory - 10 items (BFI-10) | Preparation (baseline), 1-week post experimental session and 1-month post experimental session
  The Big Five Inventory-10 (BFI-10) is a short, validated self-report instrument designed to measure the five major dimensions of personality with minimal participant burden.
  The BFI-10 is measured from 1-Disagree strongly to 5-Agree Strongly. Depending on the personality dimension a higher (e.g., openness) or lower (e.g., neuroticism) score can be better.
Behavioral Activation and Inhibition (BAI) | Preparation (baseline), 1-week post experimental session and 1-month post experimental session
  The Behavioral Inhibition System (BIS) and Behavioral Activation System (BAS) Scales are self-report measures designed to assess individual differences in sensitivity to punishment and reward, based on Gray's Reinforcement Sensitivity Theory of personality.
  The BIS/BAS is measured from 1-Strongly disagree to 4- Strongly agree. Usually balance between BIS and BAS is considered most adaptive. Neither is better or worse, universally.
Barcelona Music Reward Questionnaire (BMRQ) | Preparation (baseline), 1-week post experimental session and 1-month post experimental session.
  The Barcelona Music Reward Questionnaire (BMRQ) is a 20-item self-report scale that assesses individual differences in the sensitivity to music-induced reward across five domains: Musical Seeking, Emotion Evocation, Mood Regulation, Social Reward, and Sensory-Motor responses. Scores are summed within each domain and can also be aggregated into a global score.
  The BMRQ is measured from 1 (Completely disagree) to 5 (Completely agree). Generally a higher score is better, reflecting stronger emotional, motivational, and social responses to musical experience.
Wonder (GEMS-Wonder) | 1-day after experimental session
  Feelings of awe, amazement, transcendence in response to music
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  A higher Wonder score is strongly aligned with mystical-type experiences and positive outcomes in psilocybin research (e.g., meaning, connectedness)
Transcendence (GEMS-Transcendence) | 1-day after experimental session
  Spiritual uplift, timelessness, and "beyond-the-self" states
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  A higher Transcendence score is closely tied to beneficial mystical experiencers and long-term well-being gains.
Tenderness (GEMS-Tenderness) | 1-day after experimental session
  Warmth, empathy, affection, emotional closeness
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  A higher Tenderness score supports prosocial feelings and can lead to increased compassion and positive social outcomes.
Peacefulness (GEMS-Peacefulness) | 1-day after experimental session
  Calmness, relaxation, inner quiet.
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  A higher Peacefulness score is associated with positive acute states, reduced anxiety, and therapeutic benefit under supportive conditions.
Power (GEMS-Power) | 1-day after experimental session
  Strong, energetic, dominant feelings of drive or determination
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  Power can be positive and support motivation and agency but is not consistently linked to psilocybin outcomes; sometimes associated with intensity that can become challenging. P
Tension (GEMS-Tension) | 1-day after experimental session
  Unease, restlessness, suspense, emotional strain.
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  High Tension scores are often associated with challenging experiences and negative acute outcomes, though mild tension may precede later therapeutic insights.
Sadness (GEMS-Sadness) | 1-day after experimental session
  Unease, restlessness, suspense, emotional strain.
  The Geneva Emotional Music Scale (GEMS) is a validated, music-specific instrument designed to measure the range of emotions evoked by music.
  GEMS is scored from 0 (not at all) to 4 (extremely).
  Sadness can be cathartic and meaning-enhancing but excessive sadness may contribute to difficult experiences.
Negative-Affect Composite Factor (STAI, DASS-21, POMS Total Mood Disturbance, PANAS-Negative Affect) | Baseline; Pre-session; 1-day post-session; 1-week post-session; 1-month post-session; 1-day follow-up after the 1-month assessment.
  Composite index of negative mood/affect derived from four validated self-report measures:
  State-Trait Anxiety Inventory (STAI) : 0-3 per item; lower is better.
  Depression, Anxiety, Stress (DASS-21), 0-3 per item; lower is better.
  Profile of Mood States (POMS)-Total Mood Disturbance (TMD): 0-4 per item; lower TMD is better.
  Positive and Negative Affect Schedule (PANAS)-Negative Affect (NA) subscale: 0-4 per item; lower NA is better.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Barrett, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Psychedelics and Consciousness Research in the Behavioral Biology Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Barrett FS, Robbins H, Smooke D, Brown JL, Griffiths RR. Qualitative and Quantitative Features of Music Reported to Support Peak Mystical Experiences during Psychedelic Therapy Sessions. Front Psychol. 2017 Jul 25;8:1238. doi: 10.3389/fpsyg.2017.01238. eCollection 2017. PMID 28790944
- [Background] Barrett FS, Grimm KJ, Robins RW, Wildschut T, Sedikides C, Janata P. Music-evoked nostalgia: affect, memory, and personality. Emotion. 2010 Jun;10(3):390-403. doi: 10.1037/a0019006. PMID 20515227
- [Background] Kaelen M, Giribaldi B, Raine J, Evans L, Timmerman C, Rodriguez N, Roseman L, Feilding A, Nutt D, Carhart-Harris R. The hidden therapist: evidence for a central role of music in psychedelic therapy. Psychopharmacology (Berl). 2018 Feb;235(2):505-519. doi: 10.1007/s00213-017-4820-5. Epub 2018 Feb 2. PMID 29396616
- [Background] Golden TL, Magsamen S, Sandu CC, Lin S, Roebuck GM, Shi KM, Barrett FS. Effects of Setting on Psychedelic Experiences, Therapies, and Outcomes: A Rapid Scoping Review of the Literature. Curr Top Behav Neurosci. 2022;56:35-70. doi: 10.1007/7854_2021_298. PMID 35138585
- See also: Center for Psychedelics and Consciousness Research website — https://hopkinspsychedelic.org/musicstudy